CLINICAL TRIAL: NCT05957497
Title: Drone Biological Samples Transport Evaluation Compared to Walking in CHU CAEN NORMANDIE
Brief Title: Drone Biological Samples Transport vs Walking (DBT - Drone Biology Transport)
Acronym: DBT
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0238; 2022-A02548-35 (Registry Identifier: ID RCB)
Record Dates: First submitted 2023-03-23; First posted 2023-07-24 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-06

CONDITIONS: Healthy
Keywords: Sample transport; Drone; Pre-Analytical Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pedestrian transport: Modality of transport currently used
  Interventions: Biological: Biological samples transport and analysis
- Drone transport: Innovative modality of transport
  Interventions: Biological: Biological samples transport and analysis

INTERVENTIONS:
Biological: Biological samples transport and analysis — Biological samples transport and analysis

SUMMARY:
The transport of biological samples is a key step in the pre-analysis process in health facilities and must meet quality requirements (NF:EN:ISO 151989) to ensure that samples are transported in are transported in good conditions.

Still in the experimental stage, drone-based air transport is participating in the aeronautical revolution of the development of unmanned aircraft on board in all areas of society, including health.

This first project, led by the Biology Centre and the INNOVABIO Biological Resources Centre of the CHU de CAEN in collaboration with the company Delivrone, will allow to evaluate the feasibility in real condition of the mode of transport by drone versus transport of reference on the quality of a varied panel of medical biology examinations (biochemistry, hematology and haemostasis), on the safety of people (potentially infectious samples), on the control of the delivery time, on the control of the transport temperature (15-25°C ). The samples will be taken on 30 healthy volunteers with a total panel of 23 blood tests performed.

DETAILED DESCRIPTION:
Panel of blood tests performed on healthy volunteers samples include :

* Na, K, Cl, HC03-
* total protein
* Ca
* Creatinine, urea
* Albumine
* Bilirubin
* Liver transaminases (ALT, AST)
* Alkaline phosphatase
* GGT
* LDH
* C-reactive protein
* Complete Blood Count
* Sedimentation rate
* PT
* aPTT
* Fibrinogen
* D-Dimer

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, over 18 years old

Exclusion Criteria:

* Unhealthy volunteers previously known
* pregnant or breastfeeding woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Impact on Sodium test | 1 day
  Evaluation difference between results of Sodium (mmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Potassium test | 1 day
  Evaluation difference between results of Potassium (mmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Chlorure test | 1 day
  Evaluation difference between results of Chlorure (mmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Bicarbonate test | 1 day
  Evaluation difference between results of Bicarbonate (mmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Protein test | 1 day
  Evaluation difference between results of Protein (g/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Calcium test | 1 day
  Evaluation difference between results of Calcium (mmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Creatinin test | 1 day
  Evaluation difference between results of Creatinin (µmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Urea test | 1 day
  Evaluation difference between results of Urea (mmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Albumin test | 1 day
  Evaluation difference between results of Albumin (g/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Bilirubin test | 1 day
  Evaluation difference between results of Bilirubin (µmol/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on liver transaminase (ALT) test | 1 day
  Evaluation difference between results of liver transaminase (ALT, U/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on liver transaminase (AST) test | 1 day
  Evaluation difference between results of liver transaminase (AST, U/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on alkalin phosphatase test | 1 day
  Evaluation difference between results of alkalin phosphatase (U/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on GGT test | 1 day
  Evaluation difference between results of GGT (U/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on LDH test | 1 day
  Evaluation difference between results of LDH (U/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on C-reactive Protein test | 1 day
  Evaluation difference between results of C-reactive Protein (mg/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on red blood cells count | 1 day
  Evaluation difference between results of red blood cells (T/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on hemoglobin test | 1 day
  Evaluation difference between results of hemoglobin (g/dL) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on white blood cells count | 1 day
  Evaluation difference between results of white blood cells (G/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on neutrophil cells count | 1 day
  Evaluation difference between results of neutrophil cells (G/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on lymphocytes cells count | 1 day
  Evaluation difference between results of lymphocytes cells (G/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on platelets count | 1 day
  Evaluation difference between results of platelets (G/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on sedimentation rate test | 1 day
  Evaluation difference between results of sedimentation rate (mm) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on PT test | 1 day
  Evaluation difference between results of PT (sec and %) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on a-PTT test | 1 day
  Evaluation difference between results of a-PTT (sec) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on Fibrinogen test | 1 day
  Evaluation difference between results of Fibrinogen (g/L) after drone transport (30 samples) versus pedestrian transport (30 samples).
Impact on D-Dimer test | 1 day
  Evaluation difference between results of D-Dimer (ng/mL) after drone transport (30 samples) versus pedestrian transport (30 samples).

SECONDARY OUTCOMES:
Evaluation of the users security | 1 day
  Report accident of drone or users injuries
Evaluation of the users safety | 1 day
  Report numbers of samples broken (contamination risk) after drone transport
Temperature | 1 day
  Temperature measurement during the transport. Evaluation of the ambient temperature respect during the transport in the two conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin GILLET, MD, Study Chair — CHU CAEN NORMANDIE
Locations (1):
- Chu Caen Normandie, Caen, France